CLINICAL TRIAL: NCT02582567
Title: Effects of Supervised Exercise During Gestation on Maternal and Foetal Health Markers. The GESTAFIT Project
Brief Title: Effects of Exercise During Gestation on Maternal and Foetal Health
Acronym: GESTAFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Virginia A. Aparicio García-Molina, PhD, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: GESTAFIT
Record Dates: First submitted 2015-10-06; First posted 2015-10-21 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy
Keywords: Pregnant Women; Quality of Life; Exercise; Sleep; Fetal Research; Diet, Mediterranean; Physical Fitness; Oxidative stress; Inflammation
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gestafitos (Experimental): This is a longitudinal study developed, which is the continuation of the GESTAtion and FITness (GESTAFIT) Project. The main purpose is to evaluate the influence of a concurrent physical exercise program during pregnancy (developed under the GESTAFIT project) on the body composition, physical fitness, brain structure, and motor, cognitive, and language development of the offspring at four years of age.
  Interventions: Other: Exercise intervention; Other: Control group
- Placentraining (Experimental): This is a retrospective study which purpose is to analyse the status of placentas of women participating in the GESTAFIT project, in which a concurrent physical exercise programme was developed. This rigorous design will allow us to test our central hypothesis that exercise during pregnancy will produce greater improvements in placental metabolic pathways associated with pregnancy complications, and is associated with better pregnancy and newborn outcomes.
  Interventions: Other: Exercise intervention; Other: Control group

INTERVENTIONS:
Other: Exercise intervention — The exercise intervention will be performed in two groups so that each group will have 12-13 participants.The groups will train 3 days/week (60min per session) from the 16th week of gestation until delivery. The exercise intervention group will go through different phases of training: a) Learning phase: which will involve the intervention plan, the goals we want to work, and how we will perform it; b) Movement Learning phase: theoretical and practical sessions with the explanation of movements and ergonomic basic patterns; and c) Physical Fitness Training phase: with training sessions aimed at improving fitness and weight loss, and training sessions focused on a correct pelvic mobilization for the delivery.The intensity will be adapted during the exercise program based on the week of gestation and each pregnant heart rate. The sessions will consist of a mixed work, composed of circuits where both muscular and cardiovascular conditioning will be implemented.
Other: Control group — Usual care, not exercise.

SUMMARY:
The main objective of this project is to assess the effects of a novel and supervised exercise intervention in overweight pregnant and their newborn.

Methods/Design: The present study is a Randomized Controlled Trial. Sixty overweight pregnant interested in participate in the intervention program will be randomly assigned to either exercise (3 sessions/week), or to usual care (control) group (30 pregnant per group). The primary outcome measures are maternal weight gain, and maternal and neonatal glycaemic profile. Secondary outcomes measure are: i) body composition; ii) dietary patterns; iii) physical fitness; iv) objectively measured physical activity and sedentary behaviour; v) sleep quality; vi) mental health, quality of life and positive health; vii) haematology and biochemical analysis; viii) oxidative stress; ix) pro- and anti-inflammatory markers; x) bone health biomarkers; xi) adiposity-related proteins expression. The data will be analysed on an intention-to-treat basis and per protocol.

ELIGIBILITY:
Inclusion criteria:

* Overweight pregnant woman with a normal pregnancy course.
* Answer "no" to all questions on the PARmed-X for pregnancy*.
* To be able to walk without assistance.
* To be able to read and write enough.
* Informed consent: To be capable and willing to provide consent. *In addition, specific inclusion criteria for data analysis are: gestational age at delivery of 37-42 weeks with single foetus, spontaneous vaginal delivery or instrumental vaginal and caesarean without maternofoetal pathology (or other indication that does not involve maternofoetal risk, such as disproportion, failed induction, no foetal progression or non-cephalic presentation), newborn with appropriate weight, Apgar score>7 in the 1st and 5th minute of life, cord blood pH (normal>7.20) and normal monitoring results.

Exclusion criteria:

* Acute or terminal illness.
* Malnutrition.
* Inability to conduct tests for assessing physical fitness or exercise during pregnancy.
* Underweight, normal-weight or obesity.
* Pregnancy risk factors (such as hypertension, type 2 diabetes, etc.).
* Multiple pregnancies.
* Chromosopathy or foetal malformations.
* Uterine growth restriction.
* Foetal death.
* Upper or lower extremity fracture in the past 3 months.
* Presence of neuromuscular disease or drugs affecting neuromuscular function
* Be registered in other exercise program
* Perform more than 300 minutes of at least moderate physical activity per week
* Unwillingness to either complete the study requirements or to be randomised into control or intervention group.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity derived from the homeostatic model assessment for insulin resistance (HOMA-IR) | 34th week of gestation
  Insulin sensitivity will be derived from the homeostatic model assessment for insulin resistance (HOMA-IR), which will be calculated using the formula [fasting insulin (μIU/mL) x fasting glucose (mg/dL)]/405.
Maternal weight gain (kg) | 34th week of gestation
  Maternal weight gain will be defined as the weight change from baseline measurement to the last measurement
Neonatal insuline-glucose index | At delivery in cord blood samples
  Neonatal insulin sensitivity will be assessed through the ratio glucose/insulin.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure (mmHg) | at the 16th and 34th week of gestation
  Systolic and diastolic blood pressure (mmHg) will be measured after 5 minutes of rest, on 2 separate occasions (with 2 minutes between trials), with the person seated (Omron Health Care Europe B.V. Hoolddorp). The lowest value of the two trials will be selected for the analysis.
Resting heart rate (bpm) | at the 16th and 34th week of gestation
  Resting heart rate (bpm), will be measured after 5 minutes of rest, on 2 separate occasions (with 2 minutes between trials), with the person seated (Omron Health Care Europe B.V. Hoolddorp). The lowest value of the two trials will be selected for the analysis.
The Mediterranean Diet Score | at the 16th and 34th week of gestation
  The Mediterranean Diet Score in a version adapted to the specific needs during pregnancy for Fe, Ca and folic acid will be used to assess the adherence to the traditional Mediterranean dietary pattern.
Cardiorespiratory fitness (Vo2max) | at the 16th and 34th week of gestation
  The modified Bruce protocol will be performed to estimate maximal oxygen uptake (VO2max), and will be used as measure of cardiorespiratory fitness.
Cardiorespiratory fitness (meters in the 6-min walk test) | at the 16th and 34th week of gestation
  We perform the 6-minute walk test, which measures the maximum distance (in meters) each participant can walk in 6 minutes along a 45.7 m rectangular course.
Muscle strength (kg) | at the 16th and 34th week of gestation
  The handgrip strength test will be used as measure of strength
Flexibility (cm) | at the 16th and 34th week of gestation
  The back-scratch test will be used as measure of flexibility
Physical activity and sedentary behaviour (in minutes) | at the 16th, 24th and 34th week of gestation
  Accelerometry will be used to objectively assess physical activity and sedentary time. Women will be asked to wear a tri-axial accelerometer (ActiSleep+, Pensacola, Florida, United States) for 9 consecutive days, starting the same day they receive the monitor (e.g. participants who receive the accelerometer on Monday, will carry the device until Tuesday of the next week). Participants will be instructed to wear the accelerometer during the whole day (24 hours) on their wrist attached by an elastic belt. Time (in minutes) engaged in light, moderate, and moderate-vigorous intensity PA and sedentary time will be calculated. This accelerometer has been previously used in pregnancy with similar methodology as described in the present protocol.
Sleep behaviours (through accelerometry) | at the 16th, 24th and 34th week of gestation
  Behaviours related to sleep, such as sleep onset, sleep latency, total sleep time, number and duration of awakenings and sleep efficiency will be objectively calculated by using a triaxial accelerometer (ActiSleep+, Pensacola, Florida, United States). The data analysis of such ActiSleep accelerometry data will be carried out through its specific software (Actilife).
Pittsburgh Sleep Quality Index | at the 16th, 24th and 34th week of gestation
  It will be used to assess sleep quality and disturbances over a l-month time interval.
Insomnia Symptoms Questionnaire | at the 16th, 24th and 34th week of gestation
  The presence of symptoms of insomnia will be measured with the Insomnia Symptoms Questionnaire, validated in pregnant women.
Quality of life (Short-Form Health Survey 36) | at the 16th and 34th week of gestation
  We will use the Short-Form Health Survey 36, for assessing health-related quality of life.
Epidemiological Studies-Depression Scale questionnaire | at the 16th and 34th week of gestation
  The pregnant antenatal depression levels will be assessed by the Center for Epidemiological Studies-Depression Scale questionnaire, which is validated and widely employed in pregnancy.
State Trait Anxiety Index. | at the 16th and 34th week of gestation
  Anxiety levels will be assessed with the State Trait Anxiety Index.
The Detention of Restless Legs Syndrome questionnaire | at the 16th and 34th week of gestation
  The "Restless Legs Syndrome" largely determines the quality of life for many pregnant and is related to their levels of depression and sleep quality. The Spanish version of the Detention of Restless Legs Syndrome questionnaire will be employed to assess the presence and severity of this syndrome .
Oswestry Disability Index score | at the 16th and 34th week of gestation
  Low-back pain will be assessed with the Spanish version of the Oswestry Disability Index score
Pain Visual Analogue Scale | at the 16th and 34th week of gestation
  Low-back pain intensity will be also assessed with the Pain Visual Analogue Scale
6-item Female Sexual Function Index | at the 16th and 34th week of gestation
  The 6-item Female Sexual Function Index will be used to assess sex function. This instrument is composed of six questions: desire, arousal, lubrication, orgasm, satisfaction and pain. Each question can be scored from 0 to 5 and then summed up to provide a total score.
Positive health | at the 16th and 34th week of gestation
  "Positive health" will be evaluated through the following questionnaires:
  1. The Trait Meta-Mood Scale
  2. The Positive and Negative Affect Schedule
  3. The Satisfaction with Life Scale
  4. The 10-item Connor-Davidson Resilience Scale
Haematology | at 34th week of gestation and at delivery
  Erythrocyte count, haematocrit, haemoglobin, platelets, leukocytes and erythrocyte mean corpuscular volume will be quantified by Coulter (Brand).
Lipid profile (in mother and cord blood) | at 34th week of gestation and at delivery
  Plasma total, high-density lipoprotein and low-density lipoprotein cholesterol and triglycerides (all in mg/dL) will be assessed using an autoanalyzer (Hitachi-Roche p800, F. Hoffmann-La Roche Ltd. Switzerland)
Glycaemic profile (in mother and cord blood) | at 34th week of gestation and at delivery
  Plasma glucose, insulin and glycosylated haemoglobinwill be assessed using an autoanalyzer (Hitachi-Roche p800, F. Hoffmann-La Roche Ltd. Switzerland)
Total plasma antioxidant capacity (in mother and cord blood) | at 34th week of gestation and at delivery
  It will be measured by using commercial kit (spectrophotometry).
Plasma liposoluble antioxidants (in mother and cord blood) | at 34th week of gestation and at delivery
  Plasma vitamin E, retinol, carotene, coenzyme Q10 and coenzyme Q9 will be measured through mass spectrometry
Antioxidant enzymes activity (in mother and cord blood) | at 34th week of gestation and at delivery
  Eritrocite membrane catalase, glutathione peroxidase and superoxide dismutase enzymes will be by measured by spectrophotometry.
Carbonyl proteins (in mother and cord blood) | at 34th week of gestation and at delivery
  Measurement of carbonyl proteins will be done by using commercial kit (spectrophotometry).
Oxidative damage to lipids (in mother and cord blood) | at 34th week of gestation and at delivery
  Measurement of 4-hydroxynonenal and isoprostanes in urine and plasma and hydroperoxides in plasma and erythrocyte membrane by using commercial kits (spectrophotometry and ELISA)
Oxidative damage to DNA (in mother and cord blood) | at 34th week of gestation and at delivery
  measurement of 8-hydroxyguanosine in urine and plasma by commercial kits (ELISA).
Pro- and anti-inflammatory signal (in mother and cord blood) | at 34th week of gestation and at delivery
  Some maternal and umbilical cord plasma pro-inflammatory and anti-inflammatory cytokines (IL-1β, IL-2, IL-6, IL-8, IL-10, IFN-γ and TNF-α, IL-1ra and TNF Srii α), some adipokines (adiponectin, adipsin, resistin, PAI-active, insulin and leptin) and myokines (irisin) will be measured by the employment of Luminex xMAP technology.
Bone biomarkers (in mother and cord blood) | at 34th week of gestation and at delivery
  Various relevant biomarkers related to bone metabolism (ACTH, DKK-1, FGF-23, Osteocalcin, OPN-Osteopontin, Osteoprotegerin, PTH and SOST) will be measured with Luminex xMAP technology.
Adiposity-related proteins expression (in mother and cord blood) | At delivery
  Glucocorticoid receptor; peroxisome proliferation activated receptor (PPAR); the beta-11 hydroxysteroid dehydrogenase type I (11βHSD1), and beta-11 hydroxysteroid dehydrogenase type II (11βHSD2) will be assessed in maternal and umbilical cord blood and in oral mucosa from the mother and newborn.
  Moreover, 4 genes highly involved in foetal and postnatal development of adipose tissue have been selected; two are receptors: the Glucocorticoid receptor and the PPAR-γ, and two are metabolic enzymes: beta-11 hydroxysteroid dehydrogenase type I or 11βHSD1, and 11 beta-hydroxysteroid dehydrogenase type II or 11βHSD2. Of great importance are PPAR-γ1 and PPAR-γ2, which are generated from the same gene by alternative promoter usage and mRNA. We will measure such proteins as well as paraoxonase/arylesterase 1 (PON1) concentrations in maternal and umbilical cord plasma by Polymerase Chain Reaction and Western Blot techniques.
Anthropometry and Body Composition of the Mother and Child (Gestafitos) | 4 ± 1 years after birth
  The height of the mother and child will be recorded using a scale (Seca 22, Hamburg). A comprehensive analysis of body composition will be carried out for both the mother and child (DXA, Hologic Discovery QDR, Nasdaq). We will also record weight (Inbody R20, Biospace, Korea) as well as waist and neck circumference in both the mother and child.
Blood Pressure and Resting Heart Rate of the Mother and Child (Gestafitos) | 4 ± 1 years after birth
  Systolic and diastolic blood pressure, along with heart rate, will be measured three times after 5 minutes of rest (Omron Hoolddorp) in both mother and child.
Nutritional Status of the Mother and Child (Gestafitos) | 4 ± 1 years after birth
  A food frequency questionnaire and a Mediterranean Diet Adherence questionnaire will be administered. The use of nutritional supplements will also be recorded.
Physical Activity, Sedentary Behavior, and Sleep Quality of the Mother and Child | 4 ± 1 years after birth
  We will assess physical activity, sedentary behavior, and sleep-related behaviors (latency, efficiency, etc.) using accelerometers (ActigraphGT3X+, Pensacola, Florida, USA) worn on the wrist for nine consecutive days. Acceleration changes will be recorded in 5-second epochs for children and 60-second epochs for mothers. Data will be collected on total volume and intensity of activity (mean physical activity intensity), energy expenditure, and the number of minutes per day spent at various intensities: low (sedentary), light, moderate, vigorous, and moderate-to-vigorous. Sleep quality will also be recorded using the specific Actisleep software.
Health-Related Physical Fitness of the Child: PREFIT Battery | 4 ± 1 years after birth
  Muscular strength, cardiorespiratory fitness, balance, speed, and motor coordination-agility will be assessed using the following PREFIT battery tests: 20m shuttle run test, handgrip dynamometry, standing long jump test, one-leg balance test, and 4x10m shuttle run test, respectively. The PREFIT battery is a feasible, reliable, maximal, and valid tool to assess physical fitness in preschool-aged children.
Brain Structure, Cerebral Blood Flow, and Brain Function via Structural and Functional Magnetic Resonance Imaging (Gestafitos) | 4 ± 1 years after birth
  MRI will be conducted at the Brain, Mind and Behavior Research Center (CIMCYC) at the University of Granada. Dr. Irene Esteban-Cornejo, a team member, has coordinated the neuroimaging area of previously funded studies (e.g., the ACTIVEBRAINS project, a randomized controlled trial assessing the effect of exercise on the brain in children). She has completed two research stays at the Monash Institute of Cognitive and Clinical Neurosciences in Australia, holds a Master's degree in advanced MRI analysis, and is the first author of the first two brain articles from the ACTIVEBRAINS project, both published in the prestigious journal Neuroimage. Dr. Esteban-Cornejo has also worked with leading experts in exercise and brain health (Erickson KI, Kramer AF, and Hillman CH) at Northeastern University and the University of Pittsburgh. Dr. Erickson and neuroscientist Marina López-Solà are also part of the current project team.
Cognition (Gestafitos) | 4 ± 1 years after birth
  Three key aspects of executive function will be assessed:
  1. Cognitive Inhibition: Assessed via the Stroop test, which involves three conditions evaluating interference when identifying the ink color of words that do not match their meaning.
  2. Cognitive Flexibility: Assessed with two independent tests:
     Design Fluency Test: Consists of three progressive conditions where participants create unique designs under different rules in 60 seconds, assessing flexibility, creativity, and visual pattern generation.
     Trail Making Test: Five conditions assessing visual search speed, attention, mental flexibility, working memory, and motor function.
  3. Working Memory: Assessed with a computerized n-back task (see MRI section), which evaluates the ability to simultaneously store and process information.
  4. Intelligence: Assessed with the Kaufman Brief Intelligence Test (KBIT), which includes subtests for verbal and non-verbal intelligence.
Academic Performance (Gestafitos) | 4 ± 1 years after birth
  1. Woodcock-Muñoz III Battery: Spanish adaptation of the Woodcock-Johnson III (WJ III), composed of 22 subtests that assess language, mathematics, and science. Selected subtests will be used to assess math fluency, calculation, comprehension, and writing.
  2. School Grades: Parents will also be asked to provide the child's school grades from the academic year(s) during which the assessments take place.
  Other Motor, Cognitive, and Language Development Scales:
  1. Bayley Scales of Infant Development, Third Edition (BSID-III)
  2. Wechsler Intelligence Scale for Children
  3. BENCI Battery (Computerized Neuropsychological Assessment Battery for Children)
Genetic and Epigenetic Analyses (Gestafitos) | 4 ± 1 years after birth
  Buccal mucosa samples will be collected from children to analyze the expression of the FTO gene polymorphism rs9939609 and MC4R gene polymorphism rs17782313. DNA will be extracted from saliva using Whatmann® paper supports and organic extraction methods optimized for quality and quantity. Samples will be quantified using a NanoDrop 2000 spectrophotometer (ThermoScientific) and normalized to ~5 ng/µL before being genotyped with TaqMan probes (Applied Biosystems) on a RealTime ABI PRISM® 7900 HT. Unsuccessful samples will be amplified and sequenced using specific primers and analyzed with the 3130 HID Genetic Analyzer (Applied Biosystem). DNA and RNA will be extracted using the QIAamp DNA Mini Kit and DNeasy Blood & Tissue Kit (Qiagen), and processed with the Qiacube robot.
Oxidative stress and antioxidant defence (Placentraining) | after placental expulsion following birth
  The content in placenta of fat-soluble antioxidants (tocopherol, coenzyme Q10 and Q9 and retinol) will be analysed by HPLC, and nitric oxide and the total antioxidant capacity by the ABTS method.
  * Oxidative damage to proteins: carbonyl proteins using commercial kits (spectrophotometry).
  * Oxidative damage to lipids: 4-hydroxynonenal and isoprostanes using commercial kits (spectrophotometry and ELISA). Oxidative damage to DNA: 8-hydroxyguanosine by commercial kits (ELISA).
Expression of markers of biogenesis, autophagy, mitochondrial fusion-fission processes (Placentraining) | after placental expulsion following birth
  Changes inmitochondrial dynamics and their quality control are a key aspect to explain the observed findings.
  Therefore, using Western-blotting or RT-PCR, the mitochondrial processes of fission (Drp1, Fis1 and OPA1), fusion (Mfn1 and Mfn2), biogenesis (PGC1alpha, Tfam, Sirt1, Nrf1, Nrf2) and autophagy (PARKIN2, PINK1, Beclin-1, ATG8, ATG5, ATG12, VDAC1).
Trace and ultra-trace minerals (Placentraining) | after placental expulsion following birth
  The determination of total content of these essential (Ca, Mg, Mn, Fe, Cu, Zn, Se) or toxic elements (Hg, V, Cr, As, Cd, Pb, Ni) in placenta samples will be performed by an ICP-MS instrument (Agilent 7500, Agilent Technologies, Tokyo, Japan) fitted with a Meinhard type nebulizer (Glass Expansion, Romainmotier) and equipped with a He collision cell.
Genomic and methylation (Placentraining) | after placental expulsion following birth
  Samples will be processed as it is previously described in the "Genetic analyses section". Genomic and Methylation will be developed by pyrosequencing method. This will be developed for detection of FTO and MC4R genes. Genomic DNA from placentas will be isolated using DNeasy Blood&Tissue Kit following the recommended protocol (Qiagen N.V, Hi.GE). After checking the quality and quantity of the DNA, the promoters of the FTO and MC4R genes will be amplified by means of predesigned PyroMark CpG Assays. Region amplification using these primers will allow us to directly quantify the methylation status of the CGs within the region. First, we will amplify FTO and MC4R regions of interest by PCR using the PyroMark PCR Kit (QIAGEN N.V, Hi.GE), which enables labelling CG nucleotides susceptible of being methylated. Reaction products (one per sample and gene) will be purified and used for the sequencing reaction.
Candidate gene expression and Small RNA analysis (Placentraining) | after placental expulsion following birth
  For a better understanding of the metabolic pathways involved, we will carry out the study of candidate genes, as well as the determination of miRNAs that will allow us to establish a genotype-expression-environment relationship (with Small RNA Sequencing analysis).
  For mRNA and miRNA analysis, placental RNA will be obtained through the kit "RNeasy Mini" (Qiagen) following the manufacturer instructions. RNA integrity will be analyzed by a "RNA 6000 Nano chip" (Agilent) using a Bionalalyzer 2100 (Agilent) and the concentration will be calculated by NanoDrop 2000 (ThermoFisher Scientific).
  Predesigned TaqMan Gene Expression assays (ThermoFisher Scientific) will be used to study the expression of candidate genes: IL6, CXCL8, TNF-alpha, CSF3, BDNF; FTO, MC4R and KL klotho (KL).
Targeted and untargeted metabolomics and lipidomics analyses | after placental expulsion following birth
  Targeted metabolomics analyses will be performed using liquid chromatography coupled to mass spectrometry. Lipid species extraction will be extracted from plasma samples with MTBE. Ten μL of the extracted sample will be applied onto UPLC 1290 (Agilent Technologies, Barcelona, Spain) equipped with a reversed-phase column coupled to QTOF mass spectrometer model 6545 (Agilent Technologies, Barcelona, Spain). Data will be collected in positive and negative electrospray modes. MassHunter (Agilent Technologies, Barcelona, Spain) and R software will be used to collect, extract, align, filter and normalize the data using quality controls. Untargeted metabolomics analyses will be performed using liquid chromatography coupled to mass spectrometry. Metabolite extraction will be extracted from plasma samples with methanol.
Toxics (Placentraining) | after placental expulsion following birth
  Concentrations of free bioactive phenols will be determined by multiclass ultra-high-performance liquid chromatography-tandem mass spectrometry (UHPLC-MS/MS). The following phenols will be assessed:
  bisphenol A; parabens: methylparaben, ethylparaben, propylparaben, butylparaben; benzofenonas (BzP): BzP-1, BzP-2, BzP-3, BzP-6, BzP-8, 4-hydroxy-BzP. Concentrations of perfluoroalkyl substances in placenta will be assessed by coupling salt assisted liquid-liquid extraction with dispersive liquid-liquid microextraction and UHPLC-MS/MS. The following perfluoroalkyl substances will be measured: PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnA, PFDoA, PFTrA, PFHxS and PFOS.
Inflammatory, anti-inflammatory, vasculogenesis and angiogenesis markers (Placentraining) | after placental expulsion following birth
  We will use Luminex xMAP technology (Millipore, Darmstadt, Germany) kits to assess placenta Fractalkine, IL-1α, IL1β, IL-RA, IL-2, IL-6, IL-8, IL-10, IFN-γ, TNF-α, TNF-β, Brain-derived neurotrophic factor, Epidermal growth factor, Fibroblast growth factor 2, Granulocyte-colony stimulating factor, Granulocyte-macrophage colony-stimulating factor, Platelet-derived growth factor-AA, Monocyte chemoattractant protein-1, Vascular endothelial growth factor. For these determination we will use Human Sepsis Magnetic Bead Panel 3 Multiplex Assay (cat. No. HTH17MAG-14K).

CONTACTS AND LOCATIONS:
Locations (1):
- Pilar Cabello-Turmo, Granada, Granada, Spain

REFERENCES:
- [Derived] Marin-Jimenez N, Baena-Garcia L, Coll-Risco I, Flor-Alemany M, Castro-Pinero J, Aparicio VA. Influence of a Concurrent Exercise Training Program on Health-Related Quality of Life During Advanced Pregnancy: The GESTAFIT Project. Sports Health. 2024 Jul-Aug;16(4):518-526. doi: 10.1177/19417381231189730. Epub 2023 Jul 31. PMID 37525559
- [Derived] Aparicio VA, Baena-Garcia L, Flor-Alemany M, Martinez-Gonzalez LJ, Varela-Lopez A, Sanchez C, Quiles JL. Differences in maternal and neonatal cardiometabolic markers and placenta status by foetal sex. The GESTAFIT project. Womens Health (Lond). 2022 Jan-Dec;18:17455057221117976. doi: 10.1177/17455057221117976. PMID 35989614
- [Derived] Baena-Garcia L, Coll-Risco I, Ocon-Hernandez O, Romero-Gallardo L, Acosta-Manzano P, May L, Aparicio VA. Association of objectively measured physical fitness during pregnancy with maternal and neonatal outcomes. The GESTAFIT Project. PLoS One. 2020 Feb 18;15(2):e0229079. doi: 10.1371/journal.pone.0229079. eCollection 2020. PMID 32069319
- [Derived] Aparicio VA, Ocon O, Diaz-Castro J, Acosta-Manzano P, Coll-Risco I, Borges-Cosic M, Romero-Gallardo L, Moreno-Fernandez J, Ochoa-Herrera JJ. Influence of a Concurrent Exercise Training Program During Pregnancy on Colostrum and Mature Human Milk Inflammatory Markers: Findings From the GESTAFIT Project. J Hum Lact. 2018 Nov;34(4):789-798. doi: 10.1177/0890334418759261. Epub 2018 Mar 30. PMID 29601268
- [Derived] Aparicio VA, Ocon O, Padilla-Vinuesa C, Soriano-Maldonado A, Romero-Gallardo L, Borges-Cosic M, Coll-Risco I, Ruiz-Cabello P, Acosta-Manzano P, Estevez-Lopez F, Alvarez-Gallardo IC, Delgado-Fernandez M, Ruiz JR, Van Poppel MN, Ochoa-Herrera JJ. Effects of supervised aerobic and strength training in overweight and grade I obese pregnant women on maternal and foetal health markers: the GESTAFIT randomized controlled trial. BMC Pregnancy Childbirth. 2016 Sep 29;16(1):290. doi: 10.1186/s12884-016-1081-y. PMID 27680325